CLINICAL TRIAL: NCT03321903
Title: Tumor Oximetry Using Electron Paramagnetic Resonance (EPR) With India Ink (Using Carbon Particulates From Carlo Erba [CE])
Brief Title: EPR Tumor Oximetry With CE India Ink
Status: Terminated | Type: Observational
Why Stopped: The research team is exploring device optimization
Sponsor: Philip Schaner (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Philip Schaner, M.D., Ph.D., Associate Professor of Medicine, Geisel School of Medicine at Dartmouth, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Other Study IDs: 29880 D17008; P01CA190193 (NIH)
Record Dates: First submitted 2017-10-20; First posted 2017-10-26 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Neoplasms, Malignant; Breast Neoplasm; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Melanoma; Skin Neoplasm; Head and Neck Neoplasms
Keywords: Oxygen; Oximetry; Electron Spin Resonance Spectroscopy; Carbon; Charcoal; Radiotherapy; India Ink; EPR; ESR; Immunotherapy
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Melanoma; Skin Neoplasms; Head and Neck Neoplasms; Anthrax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — If the India ink tattoo site is surgically excised as part of standard care for the treatment of the tumor, molecular tests may be performed on the excised tissue surrounding the ink injection site to analyze for molecular biomarkers related to hypoxia, angiogenesis, and tumor growth. The tissue analysis will explore the potential for any identifying biomarkers of the tumor that predict or otherwise are associated with variation in tumor growth or responsiveness to therapy. Subjects may choose to opt of this portion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: Intraoral Squamous Cell Carcinomas: Intraoral squamous cell carcinomas that are resected and receive adjuvant radiation therapy. These patients may receive a Carlo Erba Ink injection before surgical tumor resection, after tumor resection (in the postsurgical radiation field), or in both instances. Patients whose tumor is within 5 mm of the surface will have injections of India ink into the tumor itself and measurements made in the tumor prior to surgery. Patients whose tumor is deeper than 5 mm of the surface could participate only in the measurements of the postsurgical radiation field. EPR Oximetry measurements will be made in the tumor and/or, if applicable, over the course of radiation in the postsurgical radiation field as appropriate.
  Interventions: Device: Carlo Erba Ink Injection; Other: EPR Oximetry Measurement
- 2: Cutaneous Malignant Tumors: Patients with primary cutaneous malignant tumors (including but not limited to squamous cell carcinoma, basal cell carcinoma, or melanoma) whose tumor is within 5 mm of the surface and whose treatment plan includes surgical resection and/or postsurgical radiation therapy. These patients may receive a Carlo Erba Ink injection before surgical tumor resection, after tumor resection (in the postsurgical radiation field), in both the tumor and the postsurgical radiation field, or in the tumor prior to radiation therapy. EPR Oximetry measurements will be made in the tumor and/or, if applicable, over the course of radiation in the tumor or postsurgical radiation field as appropriate.
  Interventions: Device: Carlo Erba Ink Injection; Other: EPR Oximetry Measurement
- 3: Breast Cancers: Breast cancer patients whose treatment plan includes surgical resection followed by radiation therapy. All patients who receive a surgical resection will receive a Carlo Erba Ink injection in the radiation field after sufficient healing has occurred to the area to be injected, as determined in consultation with the treating physicians, and using topical anesthetic or local anesthetic, if the patient so desires. All patients in this cohort will be expected to agree to a minimum of one EPR Oximetry measurement in the planned radiation field prior to radiation and a minimum of one measurement made over the course of radiation therapy.
  Interventions: Device: Carlo Erba Ink Injection; Other: EPR Oximetry Measurement
- 4: Other tumors: Other tumors within 5 mm of the surface, whose planned treatment includes radiotherapy of the tumor and does not include a planned resection of the tumor. As these other qualifying malignancies are expected to occur only rarely, they will be grouped into a single cohort despite potential varied histology. These patients will receive a Carlo Erba Ink injection in their tumor prior to radiation therapy. All patients in this cohort will be expected to agree to a minimum of one EPR Oximetry measurement in the planned radiation field prior to radiation and a minimum of one measurement made over the course of radiation therapy.
  Interventions: Device: Carlo Erba Ink Injection; Other: EPR Oximetry Measurement

INTERVENTIONS:
Device: Carlo Erba Ink Injection — Carlo Erba India ink is used in this study as a paramagnetic oxygen sensor that is injected into tissue, and which, when measured using EPR Oximetry, can provide sensitive, repeated, and direct measurements of tissue oxygen. Each study participant will receive at least one ink injection of 20-50µL of Carlo Erba India Ink. The ink injection will occur within 5mm of the body surface (i.e., skin or mucosa), and may be injected into tumor, postsurgical field of radiation, and/or adjacent normal tissue. Carlo Erba Ink is an aqueous suspension composed of charcoal powder, water for injection, and a suspending agent. Carlo Erba is the name of the manufacturer that supplies the charcoal.
  Other Names: Carbon particulate suspension; Charcoal suspension
Other: EPR Oximetry Measurement — An oximetry measurement visit consists of ~ 30 minutes of continuous scans of tissue oxygen in vivo, using an oxygen sensor (i.e., India ink) injected into the tumor that is noninvasively scanned using EPR oximetry. Scans, converted into measurements of pO2, characterize the current tumor oxygen level at: (1) 'steady state' (while breathing room air), 2) response to hyperoxygenation therapy (inhaling oxygen-enriched air for 10 min), and 3) response to resuming inhaling room air. EPR measurements are repeated noninvasively throughout radiation or chemotherapy, to examine changes. The minimum number of visits depends on the patient's cohort; all may have additional measurements. If the ink injection is not surgically removed, EPR oximetry measurements can be repeated indefinitely.
  Other Names: Oxygen measurement; oximetry measurement

SUMMARY:
It has been well established that malignant tumors tend to have low levels of oxygen and that tumors with very low levels of oxygen are more resistant to radiotherapy and other treatments, such as chemotherapy and immunotherapy. Previous attempts to improve response to therapy by increasing the oxygen level of tissues have had disappointing results and collectively have not led to changing clinical practice. Without a method to measure oxygen levels in tumors or the ability to monitor over time whether tumors are responding to methods to increase oxygen during therapy, clinician's reluctance to use oxygen therapy in usual practice is not surprising.

The hypothesis underlying this research is that repeated measurements of tissue oxygen levels can be used to optimize cancer therapy, including combined therapy, and to minimize normal tissue side effects or complications. Because studies have found that tumors vary both in their initial levels of oxygen and exhibit changing patterns during growth and treatment, we propose to monitor oxygen levels in tumors and their responsiveness to hyperoxygenation procedures. Such knowledge about oxygen levels in tumor tissues and their responsiveness to hyper-oxygenation could potentially be used to select subjects for particular types of treatment, or otherwise to adjust routine care for patients known to have hypoxic but unresponsive tumors in order to improve their outcomes.

The overall objectives of this study are to establish the clinical feasibility and efficacy of using in vivo electron paramagnetic resonance (EPR) oximetry-a technique related to magnetic resonance imaging (MRI)-to obtain direct and repeated measurements of clinically useful information about tumor tissue oxygenation in specific groups of subjects with the same types of tumors, and to establish the clinical feasibility and efficacy of using inhalation of enriched oxygen to gain additional clinically useful information about responsiveness of tumors to hyper-oxygenation. Two devices are used: a paramagnetic charcoal suspension (Carlo Erba India ink) and in vivo EPR oximetry to assess oxygen levels. The ink is injected and becomes permanent in the tissue at the site of injection unless removed; thereafter, the in vivo oximetry measurements are noninvasive and can be repeated indefinitely.

DETAILED DESCRIPTION:
The study design uses consecutively enrolled patients. Patients can participate as long as they are willing, fit the criteria for being assigned to a cohort, and the India ink spot remains measurable by EPR. Patients whose ink spot is resected during usual care and who do not have or are not willing to obtain additional injections will be withdrawn. Otherwise, patients can be re-measured using the previously injected ink at any time during the course of the study.

The study is split into four cohorts, with a minimum of 1-5 patients expected to be enrolled annually in each cohort, and a total of approximately 10 subjects expected for each cohort. The cohorts are defined by the type of tumor and by scenarios when our measurements will be made relative to the patient's standard therapies: 1) intraoral tumors with planned resection and adjuvant radiation therapy; 2) cutaneous malignant tumors receiving surgical resection only, receiving radiation therapy only, or receiving both surgical resection and adjuvant radiation therapy; 3) breast tumor receiving radiation therapy following surgery; and 4) other tumors receiving radiation therapy. The diagnosis for patients in all cases assumes that an eligible tumor (or the postsurgical area receiving radiation) occurs within approximately one-half centimeter of the surface, as determined by physical exam or imaging if available. All potentially eligible subjects are approached by their treating physician; those who agree to be contacted and are subsequently consented are assigned to the cohort for which they qualify. There is no randomization and no stratification within the cohorts.

Our interest in in situ tumor oxygenation relates to the clinical need to measure oxygen in tumors prior to therapy, to understand tumor oxygen dynamics over the course of therapy, and to assess the effectiveness of oxygen modulation therapy during treatment. Our interest in the postsurgical radiation field relates to the clinical need to understand whether the temporal dynamics of oxygen within the postsurgical radiation field has the potential to enhance the effectiveness of adjuvant therapies, and to understand how changes in short and long term oxygenation within the postsurgical radiation field may facilitate diminishment of late side effects from surgery and/or radiotherapy.

Following enrollment in the study, each subject will receive an initial placement of one or more geographically separate injections of India ink into the tissue of interest (i.e., tumor and/or tumor bed and/or adjacent tissue) using the established procedures for the injection of the ink. The subject is expected to agree to periodic measurements of all injection sites (unless the ink injection has been surgically removed); the subject will be told to expect six or more visits for measurements during treatment, but must agree to have at least one measurement per injection site. Each measurement will typically consist of 3 ten minute consecutive periods during which the subject initially breathes room air, then 100% oxygen delivered through a non-rebreather face mask followed by a period breathing room air.

Patients will be evaluated during clinical and oximetry appointments with respect to the presence of any adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be capable of giving informed consent or has an acceptable surrogate capable of giving consent on behalf of the subject.
2. Subject has an eligible tumor that is within 5 mm of the surface (either skin or mucosa) or has had a tumor removed with a tumor bed that is within 5 mm of the surface.

   1. Eligible tumors types:

      * Intraoral tumors: squamous cell carcinoma (SCC), melanoma;
      * Primary cutaneous tumors (including, but not limited to): SCC, basal cell carcinoma (BCC,) melanoma;
      * Breast malignancies post surgery;
      * Other tumors: any tumor within 5 mm of the surface and with planned radiation therapy.

Exclusion Criteria:

1. Previous adverse reaction to a charcoal product e.g., a local hypersensitive response from a black tattoo or from ingestion of activated charcoal
2. Previous adverse reaction to the suspending agent
3. Subject has a pacemaker that is not known to be MRI compatible
4. Subject has a non-removable implant or device with metal that is not known to be MRI compatible
5. Subject is pregnant or has a likelihood for becoming pregnant during the basic study timeframe.

Note: There is no known harm to the woman or her fetus from participating; this is precautionary only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with eligible tumors within 5mm of the surface, or that will be receiving postsurgical radiation following the resection of eligible tumors.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2019-10-27 (Actual); Study Completion 2019-10-27 (Actual)

PRIMARY OUTCOMES:
Measurement of oxygen levels in tissues in response to hyperoxic therapy | From time of ink injection to the time the ink is removed through surgical resection. This can range from days to years, or until the study's completion of enrollment, anticipated in 2020.
  This study will assess whether the addition of hyperoxic therapy (100% oxygen delivered through a non-rebreather face mask) will increase the oxygen level of a tumor or tumor bed by > 5 mm Hg using EPR oximetry. Tumor oxygen values will be reported in millimeters of mercury (mmHg).

SECONDARY OUTCOMES:
Characterize oxygen changes in tumor beds throughout the course of radiation therapy | From time of ink injection through the completion of radiation therapy; an average of 4 months.
  This outcome will measure oxygen in the post-surgical tissue throughout the course of radiation therapy using EPR oximetry. Tissue oxygen values will be reported in millimeters of mercury (mmHg).
Characterize oxygen changes in tumors throughout the course of radiation therapy | From time of ink injection through the completion of radiation therapy; an average of 4 months.
  This outcome will measure tumor tissue oxygen throughout the course of radiation therapy using EPR oximetry. Tissue oxygen values will be reported in millimeters of mercury (mmHg).
Characterize oxygen changes in tumor and tumor beds prior to radiation therapy | From time of ink injection through the completion of medical treatment for cancer; an average of 4 months.
  For those subjects receiving India ink injections in both the untreated tumor and in the post-surgical bed prior to radiation, we will examine patterns across these two 'states' in individual tumors, which can enhance our understanding of the relationship between the oxygen levels in the tumor and in the resulting tumor bed. Tissue oxygen values will be reported in millimeters of mercury (mmHg).
Characterize oxygen changes in tumor and tumor beds through the course of radiation therapy | From time of ink injection through the completion of medical treatment for cancer; an average of 6 months.
  For those subjects receiving India ink injections in both the untreated tumor and in the post-surgical bed while undergoing radiation therapy, we will examine patterns across these two 'states' in individual tumors, which can enhance our understanding of the relationship between the oxygen levels in the tumor and in the resulting tumor bed. Tissue oxygen values will be reported in millimeters of mercury (mmHg).

OTHER OUTCOMES:
Tissue Histology | Approximately 30 days post-surgical excision of the tumor
  For those subjects whose tumor is resected along with the tissue containing the India ink carbon particles as a part of their usual care, the tissue at the site of the injection will be submitted for processing with standard pathology procedures. Tissue sections spanning the injection site(s) will be evaluated for the extent and mechanism of dispersion and for the presence of acute or chronic inflammation or other tissue reaction (scar, fibrosis, capsule formation, or other). The tissue will be assessed as to whether the reaction observed is as expected for ink injections.

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Schaner, M.D., Ph.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bacic G, Liu KJ, O'Hara JA, Harris RD, Szybinski K, Goda F, Swartz HM. Oxygen tension in a murine tumor: a combined EPR and MRI study. Magn Reson Med. 1993 Nov;30(5):568-72. doi: 10.1002/mrm.1910300507. PMID 8259056
- [Background] Baudelet C, Gallez B. How does blood oxygen level-dependent (BOLD) contrast correlate with oxygen partial pressure (pO2) inside tumors? Magn Reson Med. 2002 Dec;48(6):980-6. doi: 10.1002/mrm.10318. PMID 12465107
- [Background] Brizel DM, Scully SP, Harrelson JM, Layfield LJ, Dodge RK, Charles HC, Samulski TV, Prosnitz LR, Dewhirst MW. Radiation therapy and hyperthermia improve the oxygenation of human soft tissue sarcomas. Cancer Res. 1996 Dec 1;56(23):5347-50. PMID 8968082
- [Background] Brizel DM, Sibley GS, Prosnitz LR, Scher RL, Dewhirst MW. Tumor hypoxia adversely affects the prognosis of carcinoma of the head and neck. Int J Radiat Oncol Biol Phys. 1997 May 1;38(2):285-9. doi: 10.1016/s0360-3016(97)00101-6. PMID 9226314
- [Background] Charlier N, Beghein N, Gallez B. Development and evaluation of biocompatible inks for the local measurement of oxygen using in vivo EPR. NMR Biomed. 2004 Aug;17(5):303-10. doi: 10.1002/nbm.902. PMID 15366029
- [Background] Chaplin DJ, Horsman MR. Tumor blood flow changes induced by chemical modifiers of radiation response. Int J Radiat Oncol Biol Phys. 1992;22(3):459-62. doi: 10.1016/0360-3016(92)90853-a. PMID 1735678
- [Background] Dardzinski BJ, Sotak CH. Rapid tissue oxygen tension mapping using 19F inversion-recovery echo-planar imaging of perfluoro-15-crown-5-ether. Magn Reson Med. 1994 Jul;32(1):88-97. doi: 10.1002/mrm.1910320112. PMID 8084241
- [Background] Demidenko E. Mixed models: theory and applications with R. John Wiley & Sons; 2013 Aug 26.
- [Background] Dewhirst MW, Poulson JM, Yu D, Sanders L, Lora-Michiels M, Vujaskovic Z, Jones EL, Samulski TV, Powers BE, Brizel DM, Prosnitz LR, Charles HC. Relation between pO2, 31P magnetic resonance spectroscopy parameters and treatment outcome in patients with high-grade soft tissue sarcomas treated with thermoradiotherapy. Int J Radiat Oncol Biol Phys. 2005 Feb 1;61(2):480-91. doi: 10.1016/j.ijrobp.2004.06.211. PMID 15667971
- [Background] Dunn JF, Ding S, O'Hara JA, Liu KJ, Rhodes E, Weaver JB, Swartz HM. The apparent diffusion constant measured by MRI correlates with pO2 in a RIF-1 tumor. Magn Reson Med. 1995 Oct;34(4):515-9. doi: 10.1002/mrm.1910340405. PMID 8524017
- [Background] Flood AB, Satinsky VA, Swartz HM. Comparing the Effectiveness of Methods to Measure Oxygen in Tissues for Prognosis and Treatment of Cancer. Adv Exp Med Biol. 2016;923:113-120. doi: 10.1007/978-3-319-38810-6_15. PMID 27526132
- [Background] Gallez B, Baudelet C, Jordan BF. Assessment of tumor oxygenation by electron paramagnetic resonance: principles and applications. NMR Biomed. 2004 Aug;17(5):240-62. doi: 10.1002/nbm.900. PMID 15366026
- [Background] Gallez B, Debuyst R, Dejehet F, Liu KJ, Walczak T, Goda F, Demeure R, Taper H, Swartz HM. Small particles of fusinite and carbohydrate chars coated with aqueous soluble polymers: preparation and applications for in vivo EPR oximetry. Magn Reson Med. 1998 Jul;40(1):152-9. doi: 10.1002/mrm.1910400120. PMID 9660565
- [Background] Gallez B, Swartz HM. In vivo EPR: when, how and why? NMR Biomed. 2004 Aug;17(5):223-5. doi: 10.1002/nbm.913. PMID 15366024
- [Background] Gatenby RA, Kessler HB, Rosenblum JS, Coia LR, Moldofsky PJ, Hartz WH, Broder GJ. Oxygen distribution in squamous cell carcinoma metastases and its relationship to outcome of radiation therapy. Int J Radiat Oncol Biol Phys. 1988 May;14(5):831-8. doi: 10.1016/0360-3016(88)90002-8. PMID 3360652
- [Background] Glockner JF, Swartz HM. In vivo EPR oximetry using two novel probes: fusinite and lithium phthalocyanine. Adv Exp Med Biol. 1992;317:229-34. doi: 10.1007/978-1-4615-3428-0_24. No abstract available. PMID 1337656
- [Background] Glockner JF, Norby SW, Swartz HM. Simultaneous measurement of intracellular and extracellular oxygen concentrations using a nitroxide-liposome system. Magn Reson Med. 1993 Jan;29(1):12-8. doi: 10.1002/mrm.1910290105. PMID 8380480
- [Background] Goda F, Liu KJ, Walczak T, O'Hara JA, Jiang J, Swartz HM. In vivo oximetry using EPR and India ink. Magn Reson Med. 1995 Feb;33(2):237-45. doi: 10.1002/mrm.1910330214. PMID 7707915
- [Background] Goda F, O'Hara JA, Rhodes ES, Liu KJ, Dunn JF, Bacic G, Swartz HM. Changes of oxygen tension in experimental tumors after a single dose of X-ray irradiation. Cancer Res. 1995 Jun 1;55(11):2249-52. PMID 7757972
- [Background] Goda F, O'Hara JA, Liu KJ, Rhodes ES, Dunn JF, Swartz HM. Comparisons of measurements of pO2 in tissue in vivo by EPR oximetry and microelectrodes. Adv Exp Med Biol. 1997;411:543-9. doi: 10.1007/978-1-4615-5865-1_67. No abstract available. PMID 9269471
- [Background] Haga T, Hirata H, Lesniewski P, Rychert KM, Williams BB, Flood AN, Swartz HM. L-band surface-coil resonator with voltage-control impedance-matching for EPR tooth dosimetry. Concepts in Magnetic Resonance Part B: Magnetic Resonance Engineering. 2013 Feb 1;43(1):32-40.2013).
- [Background] Hall EJ, Giaccia AJ. Radiobiology for the Radiologist. Philadelphia: JB Lippincott. 1988.
- [Background] Hees PS, Sotak CH. Assessment of changes in murine tumor oxygenation in response to nicotinamide using 19F NMR relaxometry of a perfluorocarbon emulsion. Magn Reson Med. 1993 Mar;29(3):303-10. doi: 10.1002/mrm.1910290305. PMID 8450739
- [Background] Hirata H, Walczak T, Swartz HM. Electronically tunable surface-coil-type resonator for L-band EPR spectroscopy. J Magn Reson. 2000 Jan;142(1):159-67. doi: 10.1006/jmre.1999.1927. PMID 10617447
- [Background] Hockel M, Schlenger K, Mitze M, Schaffer U, Vaupel P. Hypoxia and Radiation Response in Human Tumors. Semin Radiat Oncol. 1996 Jan;6(1):3-9. doi: 10.1053/SRAO0060003. PMID 10717157
- [Background] Hockel M, Vorndran B, Schlenger K, Baussmann E, Knapstein PG. Tumor oxygenation: a new predictive parameter in locally advanced cancer of the uterine cervix. Gynecol Oncol. 1993 Nov;51(2):141-9. doi: 10.1006/gyno.1993.1262. PMID 8276286
- [Background] Hyde JS and Subczynski, WK. Spin-label oximetry. (1989). Pp 399-425. In: Berliner LJ, Reuben J (ed). Spin Labeling: Theory and Applications. New York: Plenum Press. doi: 10.1007/978-1-4613-0743-3_8
- [Background] Islam PS, Chang C, Selmi C, Generali E, Huntley A, Teuber SS, Gershwin ME. Medical Complications of Tattoos: A Comprehensive Review. Clin Rev Allergy Immunol. 2016 Apr;50(2):273-86. doi: 10.1007/s12016-016-8532-0. PMID 26940693
- [Background] Jordan BF, Baudelet C, Gallez B. Carbon-centered radicals as oxygen sensors for in vivo electron paramagnetic resonance: screening for an optimal probe among commercially available charcoals. MAGMA. 1998 Dec;7(2):121-9. doi: 10.1007/BF02592236. PMID 9951772
- [Background] Jordan BF, Gregoire V, Demeure RJ, Sonveaux P, Feron O, O'Hara J, Vanhulle VP, Delzenne N, Gallez B. Insulin increases the sensitivity of tumors to irradiation: involvement of an increase in tumor oxygenation mediated by a nitric oxide-dependent decrease of the tumor cells oxygen consumption. Cancer Res. 2002 Jun 15;62(12):3555-61. PMID 12068004
- [Background] Jordan BF, Misson P, Demeure R, Baudelet C, Beghein N, Gallez B. Changes in tumor oxygenation/perfusion induced by the no donor, isosorbide dinitrate, in comparison with carbogen: monitoring by EPR and MRI. Int J Radiat Oncol Biol Phys. 2000 Sep 1;48(2):565-70. doi: 10.1016/s0360-3016(00)00694-5. PMID 10974477
- [Background] Jordan BF, Sonveaux P, Feron O, Gregoire V, Beghein N, Gallez B. Nitric oxide-mediated increase in tumor blood flow and oxygenation of tumors implanted in muscles stimulated by electric pulses. Int J Radiat Oncol Biol Phys. 2003 Mar 15;55(4):1066-73. doi: 10.1016/s0360-3016(02)04505-4. PMID 12605986
- [Background] Lartigau E, Randrianarivelo H, Avril MF, Margulis A, Spatz A, Eschwege F, Guichard M. Intratumoral oxygen tension in metastatic melanoma. Melanoma Res. 1997 Oct;7(5):400-6. doi: 10.1097/00008390-199710000-00006. PMID 9429223
- [Background] Lartigau E, Lusinchi A, Eschwege F, Guichard M. Tumor oxygenation: the Institut Gustave Roussy experience. In: Vaupel P, Kelleher DK (ed). Tumor hypoxia pathophysiology, clinical significance and therapeutic perspectives. Stuttgart, Germany: Wissenschaftliche Verlagsgesellschaft mbH. 1999:47-52.
- [Background] Liu KJ, Gast P, Moussavi M, Norby SW, Vahidi N, Walczak T, Wu M, Swartz HM. Lithium phthalocyanine: a probe for electron paramagnetic resonance oximetry in viable biological systems. Proc Natl Acad Sci U S A. 1993 Jun 15;90(12):5438-42. doi: 10.1073/pnas.90.12.5438. PMID 8390665
- [Background] Nakashima T, Goda F, Jiang J, Shima T, Swartz HM. Use of EPR oximetry with India ink to measure the pO2 in the liver in vivo in mice. Magn Reson Med. 1995 Dec;34(6):888-92. doi: 10.1002/mrm.1910340614. PMID 8598816
- [Background] Nilges MJ, Walczak T, Swartz HM. GHz in vivo ESR spectrometer operating with a surface probe. Phys. Med. 1989;5:195-201.
- [Background] Nordsmark M, Alsner J, Keller J, Nielsen OS, Jensen OM, Horsman MR, Overgaard J. Hypoxia in human soft tissue sarcomas: adverse impact on survival and no association with p53 mutations. Br J Cancer. 2001 Apr 20;84(8):1070-5. doi: 10.1054/bjoc.2001.1728. PMID 11308256
- [Background] Nordsmark M, Bentzen SM, Rudat V, Brizel D, Lartigau E, Stadler P, Becker A, Adam M, Molls M, Dunst J, Terris DJ, Overgaard J. Prognostic value of tumor oxygenation in 397 head and neck tumors after primary radiation therapy. An international multi-center study. Radiother Oncol. 2005 Oct;77(1):18-24. doi: 10.1016/j.radonc.2005.06.038. Epub 2005 Aug 10. PMID 16098619
- [Background] O'Hara JA, Goda F, Demidenko E, Swartz HM. Effect on regrowth delay in a murine tumor of scheduling split-dose irradiation based on direct pO2 measurements by electron paramagnetic resonance oximetry. Radiat Res. 1998 Nov;150(5):549-56. PMID 9806597
- [Background] O'Hara JA, Goda F, Liu KJ, Bacic G, Hoopes PJ, Swartz HM. The pO2 in a murine tumor after irradiation: an in vivo electron paramagnetic resonance oximetry study. Radiat Res. 1995 Nov;144(2):222-9. PMID 7480649
- [Background] O'Hara JA, Hou H, Demidenko E, Springett RJ, Khan N, Swartz HM. Simultaneous measurement of rat brain cortex PtO2 using EPR oximetry and a fluorescence fiber-optic sensor during normoxia and hyperoxia. Physiol Meas. 2005 Jun;26(3):203-13. doi: 10.1088/0967-3334/26/3/006. Epub 2005 Feb 25. PMID 15798296
- [Background] O'Hara JA, Khan N, Hou H, Wilmo CM, Demidenko E, Dunn JF, Swartz HM. Comparison of EPR oximetry and Eppendorf polarographic electrode assessments of rat brain PtO2. Physiol Meas. 2004 Dec;25(6):1413-23. doi: 10.1088/0967-3334/25/6/007. PMID 15712720
- [Background] Petryakov SV, Schreiber W, Kmiec MM, Williams BB, Swartz HM. Surface Dielectric Resonators for X-band EPR Spectroscopy. Radiat Prot Dosimetry. 2016 Dec;172(1-3):127-132. doi: 10.1093/rpd/ncw167. Epub 2016 Jul 15. PMID 27421472
- [Background] Salikhov I, Hirata H, Walczak T, Swartz HM. An improved external loop resonator for in vivo L-band EPR spectroscopy. J Magn Reson. 2003 Sep;164(1):54-9. doi: 10.1016/s1090-7807(03)00175-7. PMID 12932455
- [Background] Salikhov IK, Swartz HM. Measurement of specific absorption rate for clinical EPR at 1200 MHz. Applied Magnetic Resonance. 2005 Jun 1;29(2):287-91.
- [Background] Smirnov AI, Norby SW, Clarkson RB, Walczak T, Swartz HM. Simultaneous multi-site EPR spectroscopy in vivo. Magn Reson Med. 1993 Aug;30(2):213-20. doi: 10.1002/mrm.1910300210. PMID 8396190
- [Background] Smirnov AI, Norby SW, Walczak T, Liu KJ, Swartz HM. Physical and instrumental considerations in the use of lithium phthalocyanine for measurements of the concentration of the oxygen. J Magn Reson B. 1994 Feb;103(2):95-102. doi: 10.1006/jmrb.1994.1016. PMID 8137080
- [Background] Swartz HM. Using EPR to measure a critical but often unmeasured component of oxidative damage: oxygen. Antioxid Redox Signal. 2004 Jun;6(3):677-86. doi: 10.1089/152308604773934440. PMID 15130295
- [Background] Swartz HM. EPR Studies of Cells and Tissue. In: Foundations Of Modern EPR 1998 (pp. 451-459).
- [Background] Swartz HM. Potential Medical (Clinical) Applications of EPR: Overview & Perspectives. InIn Vivo EPR (ESR) 2003 (pp. 599-621). Springer US.
- [Background] Swartz HM, Clarkson RB. The measurement of oxygen in vivo using EPR techniques. Phys Med Biol. 1998 Jul;43(7):1957-75. doi: 10.1088/0031-9155/43/7/017. PMID 9703059
- [Background] Swartz HM, Dunn JF. Measurements of oxygen in tissues: overview and perspectives on methods. Adv Exp Med Biol. 2003;530:1-12. doi: 10.1007/978-1-4615-0075-9_1. PMID 14562699
- [Background] Swartz HM, Dunn J, Grinberg O, O'Hara J, Walczak T. What does EPR oximetry with solid particles measure--and how does this relate to other measures of PO2? Adv Exp Med Biol. 1997;428:663-70. doi: 10.1007/978-1-4615-5399-1_93. No abstract available. PMID 9500113
- [Background] Swartz HM, Halpern H. EPR studies of living animals and related model systems (in vivo EPR). InBiological magnetic resonance 2002 (pp. 367-404). Springer US.
- [Background] Swartz HM, Hou H, Khan N, Jarvis LA, Chen EY, Williams BB, Kuppusamy P. Advances in probes and methods for clinical EPR oximetry. Adv Exp Med Biol. 2014;812:73-79. doi: 10.1007/978-1-4939-0620-8_10. PMID 24729217
- [Background] Khan N, Grinberg O, Wilmot C, Kiefer H, Swartz HM. "Distant spin trapping": a method for expanding the availability of spin trapping measurements. J Biochem Biophys Methods. 2005 Feb 28;62(2):125-30. doi: 10.1016/j.jbbm.2004.10.001. Epub 2004 Nov 13. PMID 15680282
- [Background] Swartz HM, Khan N, Buckey J, Comi R, Gould L, Grinberg O, Hartford A, Hopf H, Hou H, Hug E, Iwasaki A, Lesniewski P, Salikhov I, Walczak T. Clinical applications of EPR: overview and perspectives. NMR Biomed. 2004 Aug;17(5):335-51. doi: 10.1002/nbm.911. PMID 15366033
- [Background] Swartz, HM, N. Khan, B.B. Williams, A.C. Hartford, B. Zaki, M. Ernstoff, J.C. Buckey, F.F. Gubaidullin, H. Hou, P. Lesniewski, M. Kmiec, O.Y. Grinberg, A. Sucheta, and T. Walczak, Clinical Applications of In Vivo EPR: EPR Oximetry in Treasures of Eureka, Electron Paramagnetic Resonance From Fundamental Research To Pioneering Applications & Zavoisky Award, Volume 1, Axas Publishing, New Zealand, pp. 178-179 (2009).
- [Background] Swartz HM, Iwasaki A, Walczak T, Demidenko E, Salikov I, Lesniewski P, Starewicz P, Schauer D, Romanyukha A. Measurements of clinically significant doses of ionizing radiation using non-invasive in vivo EPR spectroscopy of teeth in situ. Appl Radiat Isot. 2005 Feb;62(2):293-9. doi: 10.1016/j.apradiso.2004.08.016. PMID 15607464
- [Background] Swartz HM, Liu KJ, Goda F, Walczak T. India ink: a potential clinically applicable EPR oximetry probe. Magn Reson Med. 1994 Feb;31(2):229-32. doi: 10.1002/mrm.1910310218. PMID 8133760
- [Background] Swartz, HM, R.P. Mason, N. Hogg, B. Kalyanaraman, T. Sarna, P.M. Plonka, M. Zareb, P.L. Gutierrez, and L.J. Berliner, Free Radicals and Medicine, in Biomedical ESR a volume in the Biological Magnetic Resonance Series (S.S. Eaton, G.R. Eaton, L.J. Berliner, eds.), Kluwer Publisher (The Netherlands, New York, Boston), Chapter 3, pp. 25-74 (2004a).
- [Background] Swartz HM, Williams BB, Jarvis LA, Zaki BI, Gladstone DJ. Repeated monitoring of tumor oxygen while breathing carbogen to determine the therapeutic potential of hyperoxic therapy. Pract Radiat Oncol. 2013 Apr-Jun;3(2 Suppl 1):S23-4. doi: 10.1016/j.prro.2013.01.084. Epub 2013 Mar 25. No abstract available. PMID 24674520
- [Background] Swartz HM, Williams BB, Hou H, Khan N, Jarvis LA, Chen EY, Schaner PE, Ali A, Gallez B, Kuppusamy P, Flood AB. Direct and Repeated Clinical Measurements of pO2 for Enhancing Cancer Therapy and Other Applications. Adv Exp Med Biol. 2016;923:95-104. doi: 10.1007/978-3-319-38810-6_13. PMID 27526130
- [Background] Swartz HM, Williams BB, Zaki BI, Hartford AC, Jarvis LA, Chen EY, Comi RJ, Ernstoff MS, Hou H, Khan N, Swarts SG, Flood AB, Kuppusamy P. Clinical EPR: unique opportunities and some challenges. Acad Radiol. 2014 Feb;21(2):197-206. doi: 10.1016/j.acra.2013.10.011. PMID 24439333
- [Background] Tremper KK, Friedman AE, Levine EM, Lapin R, Camarillo D. The preoperative treatment of severely anemic patients with a perfluorochemical oxygen-transport fluid, Fluosol-DA. N Engl J Med. 1982 Jul 29;307(5):277-83. doi: 10.1056/NEJM198207293070503. PMID 7045667
- [Background] Vaeth JM. Hyperbaric oxygen and radiation therapy of cancer. Frontiers of Radiation Therapy and Oncology. 1: 195 (1968).
- [Background] Vahidi N, Clarkson RB, Liu KJ, Norby SW, Wu M, Swartz HM. In vivo and in vitro EPR oximetry with fusinite: a new coal-derived, particulate EPR probe. Magn Reson Med. 1994 Feb;31(2):139-46. doi: 10.1002/mrm.1910310207. PMID 8133749
- [Background] Vaupel P. Tumor microenvironmental physiology and its implications for radiation oncology. Semin Radiat Oncol. 2004 Jul;14(3):198-206. doi: 10.1016/j.semradonc.2004.04.008. PMID 15254862
- [Background] Vaupel P, Hockel M, Mayer A. Detection and characterization of tumor hypoxia using pO2 histography. Antioxid Redox Signal. 2007 Aug;9(8):1221-35. doi: 10.1089/ars.2007.1628. PMID 17536958
- [Background] Williams BB, Khan N, Zaki B, Hartford A, Ernstoff MS, Swartz HM. Clinical electron paramagnetic resonance (EPR) oximetry using India ink. Adv Exp Med Biol. 2010;662:149-56. doi: 10.1007/978-1-4419-1241-1_21. PMID 20204785